CLINICAL TRIAL: NCT02232503
Title: DIARET SK - Prevalence of Diabetic Retinopathy and Impact of Genetic Factors in the Development of Diabetic Retinopathy of Patients With Type 1 and 2 Diabetes Mellitus in Slovakia
Brief Title: Prevalence of DIAbetic RETinopathy and Impact of Genetic Factors in the Development of Diabetic Retinopathy of Patients With Type 1 and 2 Diabetes Mellitus in SlovaKia
Acronym: DIARET SK
Status: Completed | Type: Observational
Sponsor: Novartis Slovakia, s.r.o. (Industry)
Collaborators: Medirex Group Academy (Unknown); Slovak Technical University (Unknown); Comenius University (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002DSK01
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; Diabetes Mellitus
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — For the purpose of DNA isolation prior to genetic analysis two samples of peripheral blood will be taken. Tubes with sampled material will be stored under temperature of 2 - 8°C and in the least possible time delivered to the laboratory where DNA will be isolated. Of all the samples delivered to the laboratory, DNA will be extracted using the automated isolation method. From the second sample related to the genetic analysis also the plasma will be obtained and stored at -20°C. The DNA sample is then divided into two aliquot parts which will be stored separately for future analysis in order to decrease the risk of their impairment. DNA isolated from cells of biological material will be properly stored prior to further analysis. DNA will be archived by its freezing to -80°C, a temperature in which the characteristics are maintained for several decades.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Studied cohort — For the purpose of DNA isolation prior to genetic analysis of patients two samples of peripheral blood will be taken; first in the volume of 3.5 ml and second in the volume of 9 ml from each patient included into the study.

SUMMARY:
The aim of the study is to find out prevalence and individual stages of Diabetic Retinopathy in patients with type 1 and type 2 DM verified based on complex ophthalmologic measurements in Slovak Republic. The outcome of the project will be epidemiology survey, prevalence of diabetic retinopathy (DR) and diabetic macular edema (DME) in relation to type and duration of diabetes mellitus and risk factors. Project will also identify genetic factors linked with the diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent for epidemiological research
* Signed informed consent for genetic research
* Patients with DM - type I and II regardless of the DM duration
* All DM patients must be included regardless of presence of eye complications in patient´s anamnesis or during the examination by the diabetologist Subgroups analysis
* Patients with DM - type I and II and DM duration ≥ 20 years
* Patients with DM - type I and II and DM duration < 5 years and DR in history

Exclusion Criteria:

* Age at the time of inclusion into the <18 years
* Gestational DM or secondary-induced diabetes
* Diabetic ketoacidosis or hyperosmolar coma
* Alcohol abuse or acute alcohol intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total expected number of patients included in this survey is 5000. With the objective to guarantee non-biased patient selection sample, each screening day the pre-specified sequence of patients (5th, 10th, 15th...) will selected. If the pre-selected patient does not come for visit or does not fulfill the inclusion criteria or does not want to sign the informed consent the next patient is asked to participate in the research. We plan to enroll 4500 patients using this non-biased method.
  The weakness of the non-biased random selection is that the less frequent groups of patients will not have enough subjects for the proper statistical analysis. To correct for this effect pool of 500 patients is reserved for special subgroups. Pre-defined subgroups are:
  1. patients with DM duration more 20 years
  2. patients with DM duration less than 5 years already with DR in history All patients from these subgroups will be asked to participate in this project regardless of the pre-specified order.
Sampling Method: Probability Sample
Enrollment: 4011 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The prevalence of diabetic retinopathy as the proportion of patients with DR (any stage) in a given subgroup according to DM duration | participants screened each working day within 8 working hours during a 6 months period in selected diabetology centers according to protocol criteria
  The results will be accompanied by Wald 95% confidence intervals. The combined prevalence results from more subgroups will be evaluated using weighted average using the best available epidemiology data.

SECONDARY OUTCOMES:
Evaluate the prevalence and individual stages of Diabetic Retinopathy in patients with type 1 and type 2 DM verified based on complex ophthalmologic measurements | participants screened each working day within 8 working hours during a 6 months period in selected diabetology centers according to protocol criteria
  The calculation of prevalence for each stage of DR will be analyzed using the same methods as for the total DR prevalence.
Evaluate the prevalence and individual stages of Diabetic Macular Edema (DME) in patients with type 1 and type 2 DM verified based on complex ophthalmologic measurements | participants screened each working day within 8 working hours during a 6 months period in selected diabetology centers according to protocol criteria
  The calculation of prevalence for each stage of DME will be analyzed using the same methods as for the total DR prevalence
Evaluate the impact of risk factors on the prevalence of Diabetic Retinopathy and Diabetic Macular Edema | participants screened each working day within 8 working hours during a 6 months period in selected diabetology centers according to protocol criteria
  The analysis will be realized using multivariate logistics regression. The output of the analysis will be the impact statistical significance of the individual risk factors represented by odds ratio for each risk parameter accompanied with statistical significance and corresponding confidence interval. The risk factors will be at least: age, gender, ethnicity, DM duration since diagnosis, glycemic control and diabetes management based on the average HbA1c of all measurements in the last 12 months, presence of nephropathy, malignancies and BMI.
  Age, DM duration since diagnosis, diabetes control based on the average HbA1c of all measurements in the last 12 months and BMI will be assessed as continuous covariates whereas gender, nationality, presence of nephropathy and malignancies will be considered as categorical variables.

OTHER OUTCOMES:
Epidemiological characteristics of patients with Diabetes Mellitus and with Diabetic Retinopathy in terms of demographic structure, treatment and control of DM and the presence of other microvascular and ophthalmologic complications | participants screened each working day within 8 working hours during a 6 months period in selected diabetology centers according to protocol criteria
  The patient characteristics will be described as by standard methods of descriptive statistics - N, %, mean, media, min, max, SD and where necessary accompanied by the histogram or contingence table.
Evaluate the impact of diabetic retinopathy and diabetes mellitus on the Quality Of Life as measured by NEI-VFQ25 questionnaires | participants examined each working day within selected working hours during a 6 months period in selected ophthalmology centers according to protocol criteria
  The impact of DR and DME on the quality of life in case of patients with DM will be realized using ANCOVA method where QoL will be evaluated as the continuous variable. The multivariate analysis will include all relevant patient characteristics including visual acuity, age and gender of the patient. These characteristics will serve as covariates to correct for the difference in characteristics of patient with/without DR.
Investigate DNA polymorphisms and phenotypic features correlating with the development of DR in patients with extreme phenotypes. | DNA analysis during 7 months post study screening period
  Genetic analysis is primarily exploratory in nature, does not test the hypothesis previously postulated and formal calculation of sample size can not be determined. In combination with accurately determined ocular and diabetic history is sample size above standard within typical publications of the topic.
The analysis of mitochondrial DNA haplotypes in pre-defined patient groups | DNA analysis during 7 months post study screening period
  Basic statistical analysis will include binary logistic regression (OR, 95% CI) and Fisher test. This method evaluates the statistical significance for the increase or decrease in the risk of DR for easy single nucleotide polymorphisms (SNPs) in in mitochondrial DNA (mtDNA), their combinations - DNA haplotypes, haplogroups and their clusters and thus identifies possible genetic factors involved in the study disease.
The identification of patients with monogenic DM by biomarkers (hsCRP) | DNA analysis during 7 months post study screening period
  Calculation of prevalence HNF1A-MODY in a wide Slovak population with diabetes using biomarker hsCRP.
  Comparison of the severity of retinopathy in mutation carriers of HNF1A-MODY and type 2 diabetes / type 1 diabetes patients in the specified data set.
Identification of patients with extreme phenotypes and family history of DM with eye complications | DNA analysis during 7 months post study screening period

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Buckova, M.D., Study Director — Novartis Slovakia; Peter Carnogursky, MSc., Study Director — Novartis Slovakia, s.r.o.; Svetlana Sefcikova, MD, Study Director — Novartis Slovakia, s.r.o.; Pavol Tison, MD, Study Director — Novartis Slovakia, s.r.o.; Iveta Tvrda, MD, Study Director — Novartis Slovakia, s.r.o.; Daniela Gasperikova, MSc., PhD., Study Director — Novartis Slovakia, s.r.o.; Ivana Hojsikova, RNDr., Study Director — Medirex Group Academy; Ludevit Kadasi, RNDr., DrSc., Study Director — Comenius University; Iwar Klimes, Prof., MD, DrSc., Study Director — Novartis Slovakia, s.r.o.; Peter Jackuliak, MD, Principal Investigator — University Hospital Bratislava; Vladimir Krasnik, MD PhD., Principal Investigator — University Hospital Bratislava; Emil Martinka, MD, PhD., Principal Investigator — National Institute for Endocrinology and Diabetology; Marian Mokan, Prof. MD DrSc., Principal Investigator — Jesenius University Martin; Zuzana Nemethyova, MD, Principal Investigator — Diabetology Dispensary Bratislava; Marta Ondrejkova, MD PhD., Principal Investigator — F.D. Roosevelt Hospital Banska Bystrica; Jana Stefanickova, MD, Principal Investigator — University Hospital Bratislava